CLINICAL TRIAL: NCT03566862
Title: Audio Technology To Detect Lung Cancer Earlier
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of the West of Scotland (Other); King's College Hospital NHS Trust (Other); Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: GN16ON719
Record Dates: First submitted 2018-05-15; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Lung Neoplasms; Cough
MeSH Terms: conditions — Lung Neoplasms; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Lung cancer: Individuals with confirmed diagnosis of lung cancer including disease in the lungs and an active cough.
  Interventions: Diagnostic Test: Leicester Cough Monitor (LCM)
- COPD: Individuals with a confirmed diagnosis of COPD according to established criteria.
  Interventions: Diagnostic Test: Leicester Cough Monitor (LCM)
- Other (non-COPD) chronic lung disease: Individuals with a confirmed diagnosis of non-COPD chronic lung disease (e.g. pulmonary fibrosis, asthma).
  Interventions: Diagnostic Test: Leicester Cough Monitor (LCM)
- Normal smokers: Individuals who have presented with cough but who appear to have 'healthy' lungs (i.e. COPD, other chronic lung disease and lung cancer have been excluded after clinical assessment).
  Interventions: Diagnostic Test: Leicester Cough Monitor (LCM)

INTERVENTIONS:
Diagnostic Test: Leicester Cough Monitor (LCM) — The Leicester Monitoring Cough (LCM) kit includes a digital flash voice recorder (Sony ICD-PX333), aA clip-on lapel microphone (Philips LFH9173) and a small carry/travel waist bag.

SUMMARY:
A cross-sectional study of prospectively collected cough audio recordings using spectral analysis.

DETAILED DESCRIPTION:
In the UK lung cancer is the leading cause of cancer death, also, UK survival rates are poorer compared to other European countries. Lung cancer is plagued by late presentation; 70% present with advanced incurable disease and a third die within 90 days of diagnosis. As such, there is a clear and urgent need to achieve earlier diagnosis of lung cancer. Symptomatic presentation is the most common route to lung cancer diagnosis and symptoms may be present for many months before diagnosis, even in early stage disease. The most common (68%) presenting symptom is cough. Unfortunately cough is also common with other illnesses. Furthermore, a high proportion of those at high-risk of lung cancer have pre-existing cough or respiratory disease (e.g. ex- or current- smokers, patients with chronic obstructive pulmonary disease (COPD)). Cough sounds are known to vary according to underlying lung pathology and could therefore have diagnostic value. Potentially, there may be unique cough and/or respiratory sounds or patterns associated with lung cancer that are not detectable by the human audio spectrum. Identification of a tool that accurately discriminates lung cancer cough could be pivotal.

This is a prospective cross-sectional study that will involve subjective analysis of spectrograms of cough recorded from individuals with "normal" lungs, individuals at high-risk for lung cancer (COPD and other chronic lung diseases) and individuals with lung cancer. 24 hour ambulatory audio recordings will be prospectively collected from patients attending respiratory medicine clinics at Queen Elizabeth University Hospital (QEUH), Glasgow. Participants will be given a free-field lapel microphone and mp3 recorder for 24h. The Leicester Cough Monitor (LCM) will be used to extract the cough sounds from the 24h recordings. The LCM is an automated cough detection system that was developed by Dr Surinder Birring (Kings College Hospital). It uses an algorithm to automatically identify cough sounds from audio recordings, which is then able to provide data on cough frequency. As part of this process, the LCM splices out 1 second sound clips for all parts of the audio recordings that are identified as being (i) a cough sound or (ii) a non-cough sound.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and above and who are either:
* "Normal Smokers" - individuals who have presented with cough but who appear to have 'healthy' lungs (i.e. COPD, other chronic lung disease and lung cancer have been excluded after clinical assessment);
* "COPD" - individuals with a confirmed diagnosis of COPD according to established criteria;
* "Other (non-COPD) chronic lung disease" - individuals with a confirmed diagnosis of non-COPD chronic lung disease (e.g. pulmonary fibrosis, asthma);
* "Lung cancer" - individuals with confirmed diagnosis of lung cancer including disease in the lungs and an active cough

Exclusion Criteria:

* Participants with an active or recent lung infection, as defined by either the production of purulent sputum associated with systemic symptoms or fever, and/or the receipt of antibiotics for lung infection or acute exacerbation over the 2 weeks preceding the date of consent
* Participants who are unable to provide informed consent
* Participants who are receiving/have previously received radiotherapy to the lungs
* Participants who are currently receiving chemotherapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants for all 4 cohorts will be identified by the CI and associated research team by screening patients who attend respiratory clinics at QEUH with suspected lung cancer (for the "Normal Smokers" and Lung Cancer cohorts) and other established respiratory diseases (for the COPD and Other (non-COPD) chronic lung disease cohorts). Individuals will be recruited by the QEUH research nurse or CI when they attend the relevant outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Spectral centroid (Hz) measurement | 12 months
  Spectral centroid (Hz) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples

SECONDARY OUTCOMES:
Spectral bandwith (Hz) measurement | 12 months
  Spectral bandwith (Hz) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral crest factor (Hz) measurement | 12 months
  Spectral crest factor (Hz) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral flatness (adimensional) measurement | 12 months
  Spectral flatness (adimensional) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral flux (Watts²) measurement | 12 months
  Spectral flux (Watts²) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral roll-off (Hz) measurement | 12 months
  Spectral roll-off (Hz) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Ratio f50 vs f90 (adimensional) measurement | 12 months
  Ratio f50 vs f90 (adimensional) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral peak entropy (adimensional measurement) | 12 months
  Spectral peak entropy (adimensional measurement) of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral Renyi entropy (adimensional) measurement | 12 months
  Spectral Renyi entropy (adimensional) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral kurtosis (adimensional) measurement | 12 months
  Spectral kurtosis (adimensional) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral skewness (adimensional) measurement | 12 months
  Spectral skewness (adimensional) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples
Spectral entropy (adimensional) measurement | 12 months
  Spectral entropy (adimensional) measurement of cough sounds to ascertain any similarities or differences in spectral characteristics between samples

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Blyth, MD, Principal Investigator — NHSGG&C
Locations (1):
- Queen Elizabeth University Hospital Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No